CLINICAL TRIAL: NCT00902161
Title: A Double-Blind, Randomized, Placebo-Controlled, Single-Dose Crossover Study to Assess the Safety and Tolerability of MK0893 Coadministered With Propranolol Hydrochloride in Patients With Type 2 Diabetes
Brief Title: A Single-Dose Crossover Study of MK0893 in Patients With Type 2 Diabetes (0893-019 AM4)(COMPLETED)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 0893-019; 2009_592
Record Dates: First submitted 2009-05-13; First posted 2009-05-15 (Estimated); Results first posted 2012-05-08 (Estimated); Last update posted 2015-07-03 (Estimated); Status verified 2015-06

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — N-((4-(1-(3-(3,5-dichlorophenyl)-5-(6-methoxynaphthalen-2-yl)-1H-pyrazol-1-yl)ethyl)phenyl)carbonyl)-beta-alanine; Propranolol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Propanolol + Placebo > Propanolol + MK0893 (Experimental): Participants received propanolol for 7 weeks. On Day -1 of Period 1 (Study Visit 6), single dose MK0893-matched placebo was added and propanolol was continued. After Period 1, participants underwent a 3-week wash-out while continuing to receive propanolol. Following the washout, participants were treated with a single dose of MK0893 on Day 21 (Visit 8).
  Interventions: Drug: MK0893; Drug: MK0893-matched Placebo; Drug: Propranolol Hydrochloride (HCL)
- Propanolol + MK0893 > Propanolol + Placebo (Placebo Comparator): Participants received propanolol for 7 weeks. On Day -1 of Period 1 (Study Visit 6), single dose MK0893 was added and propanolol was continued. After Period 1, participants underwent a 3-week wash-out while continuing to receive propanolol. Following the washout, participants were treated with a single dose of MK0893-matched placebo on Day 21 (Visit 8).
  Interventions: Drug: MK0893; Drug: MK0893-matched Placebo; Drug: Propranolol Hydrochloride (HCL)

INTERVENTIONS:
Drug: MK0893 — Single dose of MK0893 1000 mg (ten 100 mg tablets)
Drug: MK0893-matched Placebo — Single dose of placebo to MK0893 (ten tablets)
Drug: Propranolol Hydrochloride (HCL) — Propranolol tablets titrated up to 80 mg three times daily over a four week period. Total treatment was approximately 7 weeks.

SUMMARY:
This study will assess the effect of combined treatment with MK0893 plus propranolol versus placebo plus propranolol on hypoglycemia.

ELIGIBILITY:
Inclusion Criteria:

* Participant has Type 2 Diabetes (T2DM)
* Participant is either: Not on an oral antihyperglycemic medication for at least 6 weeks; on a single oral antihyperglycemic medication that is not a peroxisome proliferator-activated gamma (PPAR-gamma) agonist (e.g. Avandia); OR on a combination of no more than two antihyperglycemic medications that are not PPAR-gamma) agonists
* Participant has not received insulin for at least 6 months
* Participant has not been treated with a PPAR-gamma agonist for at least 12 weeks
* Participant has been a nonsmoker for at least 6 months
* Female participants who are non-pregnant and highly unlikely to conceive due to surgical sterilization, post-menopausal status, not heterosexually active, or willing to use 2 birth control methods

Exclusion Criteria:

* Participant has a history of stroke, seizures, or neurological disorders
* Participant cannot tolerate insulin or propranolol
* Participant has a history of asthma, emphysema or chronic bronchitis
* Participant is on a weight loss program that is not in the maintenance phase or has been treated with a weight loss medication within 8 weeks of screening
* Participant is on or may require treatment with drugs that affect the immune system or with corticosteroids
* Participant has a history of heart failure or coronary artery disease
* Participant has a history of uncontrolled high blood pressure
* Participant is Human Immunodeficiency (HIV), hepatitis B or hepatitis C positive
* Participant has a history of Type 1 diabetes
* Participant has a history of hypoglycemia unawareness documented by a blood glucose concentration < 55 mg/dL (3.1 mol/L) without symptoms of hypoglycemia.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2009-05; Primary Completion 2009-10 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

RESULTS

PARTICIPANT FLOW:
Groups:
- Propanolol + MK0893 / Propanolol + Placebo: After a 4 week wash-out period with a 4-week propanolol run-on, single dose MK0893 was added on Day -1 of Period 1 (Study Visit 6) and propanolol was continued. After Period 1, participants underwent a 3-week wash-out while continuing to receive propanolol alone. Following the washout, participants were treated with a single dose of MK0893-matched placebo on Day 21 (Visit 8) while continuing on propanolol.
- Propanolol + Placebo / Propanolol + MK0893: After a 4 week wash-out period with a 4-week propanolol run-on, MK0893-matched placebo was added on Day -1 of Period 1 (Study Visit 6) and propanolol was continued. After Period 1, participants underwent a 3-week wash-out while continuing to receive propanolol alone. Following the washout, participants were treated with a single dose of MK0893 on Day 21 (Visit 8) while continuing on propanolol.
- Propanolol Alone: Participants received treatment with propanolol alone during a 4 week run-on before the 1st clamp procedure at Visit 6, and during a 3 week washout between clamp procedures at Visits 6 (Period 1) and 8 (Period 2). Overall, participants were treated with propranolol for approximately 7 weeks (from propranol titration through Visit 8 clamp procedures).
Period: Pre-study Washout/Propanolol Run-in
Arm/Group | Propanolol + MK0893 / Propanolol + Placebo | Propanolol + Placebo / Propanolol + MK0893 | Propanolol Alone
Started | 0 | 0 | 22
Completed | 0 | 0 | 22
Not Completed | 0 | 0 | 0
Period: Period 1
Arm/Group | Propanolol + MK0893 / Propanolol + Placebo | Propanolol + Placebo / Propanolol + MK0893 | Propanolol Alone
Started | 12 | 10 | 0
Completed | 12 | 10 | 0
Not Completed | 0 | 0 | 0
Period: Post-clamp Washout
Arm/Group | Propanolol + MK0893 / Propanolol + Placebo | Propanolol + Placebo / Propanolol + MK0893 | Propanolol Alone
Started | 0 | 0 | 22
Completed | 0 | 0 | 22 (2 participants discontinued washout and were replaced; 1 due to an AE and 1 due to lack of efficacy)
Not Completed | 0 | 0 | 0
Period: Period 2
Arm/Group | Propanolol + MK0893 / Propanolol + Placebo | Propanolol + Placebo / Propanolol + MK0893 | Propanolol Alone
Started | 8 | 9 | 0
Completed | 8 (2 participants discontinued and were replaced; 1 due to protocol deviation and 1 withdrew consent) | 9 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- MK0893 + Propanolol: Participants received a single dose of MK0893 added to a background of propanolol at either Visit 6 (Day -1) or Visit 8 (Day 21).
- Placebo + Propanolol: Participants received a single dose of MK0893-matched placebo added to a background of propanolol at either Visit 6 (Day -1) or Visit 8 (Day 21).
- Total: Total of all reporting groups
Arm/Group | MK0893 + Propanolol | Placebo + Propanolol | Total
Number analyzed (Participants) | 12 | 10 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.3 (5.66) | 48.5 (6.88) | 50.0 (6.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 10 | 6 | 16

OUTCOME MEASURES:

1. Primary Outcome: Recovery Time (Rt[65] From Insulin-induced Hypoglycemia
Description: Rt(65) defined as the time to recover from hypoglycemia (blood glucose level of 50 mg/dL) to an arterialized venous blood glucose of 65 mg/dL. At t= -60 minutes on the morning of Day 1 (Visit 6) or Day 22 (Visit 8), a hypoglycemic clamp was used via an increased insulin infusion rate to achieve blood glucose concentrations of 50 mg/dL (2.8 mmol/L) within ~30-90 minutes. At the end of the 30-minute hypoglycemic clamp interval, insulin and glucose infusions were terminated, and the time to recover from hypoglycemia to 65 mg/dL Rt(65) was determined. Rt(65) was followed up to 270 minutes
Time Frame: From the time of hypoglycemic clamp (t=0 minutes) through 270 minutes
Population: 21 participants who received MK0893 + Propanolol while on study had data available, and 17 participants who received Placebo + Propanolol while on study had data available
Measure: Least Squares Mean (95% Confidence Interval); unit: minutes
Groups:
- Placebo + Propanolol: Participants received a single dose of MK0893 added to a background of propanolol at either Visit 6 (Day -1) or Visit 8 (Day 21).
Arm/Group | MK0893 + Propanolol | Placebo + Propanolol
Number analyzed (Participants) | 21 | 17
minutes | 103 [88 to 118] | 71 [55 to 88]
Statistical Analysis 1: Comparison: MK0893 + Propanolol vs Placebo + Propanolol; The p-value is for testing the null hypothesis that the difference on Rt(65) between the [MK-0893 1g + Propranolol] vs. [PBO + Propranolol] >=60 min. If p-value < 0.05, then the null hypothesis is rejected at the significance level of 0.05, thus supporting the primary hypothesis that the treatment difference is less than 60 minutes; Test type: Superiority or Other; p = 0.005, A linear mixed effect (LME) model — There was only 1 primary hypothesis, so no multiplicity adjustment was required; Least Squared Mean Treatment Difference = 32, 95% CI 2-sided [15 to 49]

2. Secondary Outcome: Maximum Plasma Concentration (Cmax) and Concentration Average Over 8-12 Hours (C[Ave] 8-12 hr) Post Single Dose MK0893
Description: Cmax was the maximum or "peak" concentration of MK0893 observed after its administration.
  Approximate C(ave 8-12) was the MK0893 concentration average over 8-12 hours post-dose and was computed as the Area Under the Curve over 8-12 hours post-dose (AUC [8-12]) ÷ 4
Time Frame: From time of MK0893 administration through 24 hours post-dose
Population: Data from the first 15 participants who completed the study were used for the pharmacokinetic analysis.
Measure: Mean (Standard Deviation); unit: uM
Groups:
- MK0893: Participants received a single dose of MK0893 added to a background of propanolol at either Visit 6 (Day -1) or Visit 8 (Day 21).
Arm/Group | MK0893
Number analyzed (Participants) | 15
uM
  Cmax | 29.18 (6.51)
  C(ave) 8-12hr | 26.75 (6.04)

3. Secondary Outcome: Plasma Concentration at 32 Hours (C[32hr]) Post Single Dose MK0893
Description: Plasma concentration of single dose MK0893 was measured from time of administration to 24 hours post-dose and extrapolated out to 32 hours post-dose using the plasma concentration vs. time curve
Time Frame: From time of MK0893 administration through estimated 32 hours post-dose
Population: Data from the first 15 participants who completed the study were used for the pharmacokinetic analysis.
Measure: Mean (Standard Deviation); unit: nM
Arm/Group | MK0893 + Propanolol
Number analyzed (Participants) | 15
nM | 23.69 (4.86)

4. Secondary Outcome: Number of Participants With An Adverse Event (AE)
Description: An AE was defined as any unfavorable and unintended change in the
  structure, function, or chemistry of the body temporally associated with the use of the Sponsor's product, whether or not considered related to the use of the product. This also included any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition which is temporally associated with the use of the Sponsor's product.
Time Frame: From time of administration of study treatment through end of Post-Study (up to 21 days after administration of last dose of study treatment).
Population: All treated participants
Measure: Number; unit: participants
Groups:
- Propanolol Alone: Participants received treatment with propanolol alone during a 4 week washout before the 1st clamp procedure at Visit 6, and during a 3 week washout between clamp procedures at Visits 6 (Period 1) and 8 (Period 2). Overall, participants were treated with propranolol for approximately 7 weeks (from propranolol titration through Visit 8 clamp procedures).
Arm/Group | MK0893 + Propanolol | Placebo + Propanolol | Propanolol Alone
Number analyzed (Participants) | 22 | 22 | 22
participants | 10 | 4 | 9

5. Secondary Outcome: Number of Participants Who Discontinued Study Treatment Due To AEs
Description: as for outcome 4
Time Frame: From time of first administration of study treatment to time of last administration of study treatment (up to Day 21)
Population: All treated participants
Measure: Number; unit: participants
Arm/Group | MK0893 + Propanolol | Placebo + Propanolol | Propanolol Alone
Number analyzed (Participants) | 22 | 22 | 22
participants | 1 | 0 | 0

ADVERSE EVENTS:
Arm/Group | MK0893 + Propanolol | Placebo + Propanolol | Propanolol Alone
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 10/22 | 4/22 | 9/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK0893 + Propanolol (N=22) | Placebo + Propanolol (N=22) | Propanolol Alone (N=22)
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 0 (0)
Arrhythmia Supraventricular (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Vision Blurred (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Chest Discomfort (General disorders) | 0 (0) | 0 (0) | 1 (1)
Chest Pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 3 (3)
Feeling Hot (General disorders) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis Viral (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Wrist Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Haematocrit Decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Haemoglobin Decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Joint Effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness Postural (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 0 (0) | 3 (3)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The SPONSOR must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the SPONSOR as confidential must be deleted prior to submission. SPONSOR review can be expedited to meet publication guidelines.